CLINICAL TRIAL: NCT00959998
Title: Acupressure for Post-Treatment Cancer Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10915
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Fatigue
Keywords: Persistent Cancer-Related Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Relaxation acupressure (Active Comparator)
  Interventions: Other: Self-administered Acupressure
- High Intensity Stimulating Acupressure (Experimental)
  Interventions: Other: Self-administered Acupressure
- Low Intensity Stimulating Acupressure (Experimental)
  Interventions: Other: Self-administered Acupressure

INTERVENTIONS:
Other: Self-administered Acupressure

SUMMARY:
Persistent cancer related fatigue (PCRF) is a common symptom experienced by many cancer survivors, which may last for as long as 10 years following treatment. PCRF is currently under diagnosed, with between 20% to >60% of survivors experiencing this symptom. Currently there are few effective treatment options for these patients. Acupressure offers a potential low-toxicity self-administered treatment option to treat PCRF.

The investigators performed a pilot randomized single-blinded controlled trial of acupressure in cancer survivors experiencing moderate to severe PCRF. Potential participants were excluded if they had other causes of fatigue such as anemia, malnutrition, or chronic fatigue syndrome. Participants were randomized to one of three treatment groups: 1. relaxation acupressure (RA), 2. high intensity stimulatory acupressure (HIS), and 3. low intensity stimulatory acupressure (LIS). Participants performed acupressure for 12 weeks between 3 to 14 times per week depending on group. Fatigue was measured with the Brief Fatigue Inventory (BFI). Secondary outcomes included beliefs and expectations, assessment of blinding, compliance to treatment, demographics, and clinical parameters. The effect of group on BFI was assessed with ANOVA and linear regression. Correlations were also made between compliance and change in BFI.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 years of age and older
* A diagnosis of cancer, except for squamous and basal cell carcinomas, who had completed their cancer-related treatments at least 12 weeks prior (except for on-going hormone therapy, which must have been initiated at least three weeks prior to enrollment
* To have a complaint of persistent, moderate to severe fatigue despite standard treatment [defined as > 4 on the Brief Fatigue Inventory (BFI)]
* To maintain their typical dietary patterns, especially the use of caffeinated beverages throughout the study,

  * To be disease free and be acupuncture and acupressure naïve

Exclusion Criteria:

* Diagnosed with anemia [defined as hemoglobin levels < 12 gm/dl] or receiving treatment for anemia
* Have any comorbidities likely to cause significant fatigue (i.e., moderate to severe heart failure, hypothyroidism) either currently or before cancer diagnosis
* Have problems with easy or spontaneous bruising from any cause, e.g. bleeding disorders
* Have nutritional deficiencies [defined by albumin levels < 35 g/liter]
* Have a diagnosis of depression and are not receiving active successful treatment for depression or have a HADS depression score of ≥ 11had a diagnosis of depression and are not receiving active successful treatment for depression or have a HADS depression score of ≥ 11
* Have a thyroid disorder, defined as either thyroid stimulating hormone or free T4 lower than the normal range or greater than 2xs the upper range
* Have an anticipated survival rate of less than 6 months
* Have an initiation, a cessation or change of dose (up to three weeks prior to the study's start) of any chronic medications or dietary supplements or any planned change of chronic medications or dietary supplements during the study
* and are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To examine the effect of two intensities of self-administered stimulating acupressure compared to self-administered relaxation acupressure on severity of chronic fatigue in people diagnosed with cancer who had completed all cancer therapies | Once per week for 13 weeks

SECONDARY OUTCOMES:
Secondary objects were to evaluate the safety, tolerability, adherence, blinding and beliefs/expectation of participants of the three acupressure treatments

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States